CLINICAL TRIAL: NCT05951374
Title: Madany Triangle; a New Era of Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, Sarah Magdy Abdelmohsen, Lecturer, Aswan University Hospital
Other Study IDs: AswanUH6
Record Dates: First submitted 2023-06-19; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Laparoscopic Cholecystectomy; Cholecystitis; Gallstone
Keywords: Safe Cholecystectomy,; critical view of safety.
MeSH Terms: conditions — Cholecystitis; Gallstones

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Madany triangle — After dissection of the proximal part of the gallbladder from its bed and scarification of the cystic artery and its branches, the traction applied to the Hartman pouch created an angle between the skeletonized cystic duct and the skeletonized posterior surface of the GB (Fig. 3).
  Also, this traction creates a dynamic triangle visualized from both the left and right sides according to the traction applied to the Hartman pouch to the right or left and the direction of the angled scope of the camera lens. From the left-side view, when right traction is applied to the Hartman pouch, it is bound laterally by the skeletonized proximal part of the cystic duct. Superiorly, it is bound by the posterior surface of the proximal part of the skeletonized gallbladder. It was bounded medially by an imaginary line between a point at the junction of the cystic duct with the CBD and a point at the anterior end of the dissected cystic plate (the Madany triangle)

SUMMARY:
Laparoscopic cholecystectomy has an increased incidence of extrahepatic biliary injury or bleeding. The common hepatic duct is on the medial border of the Calot triangle and at risk of injury. So, The investigators describe a new safety triangle with a more critical view of safety that is far from dangerous.

Retrospectively, from December 2019 until March 2023, the investigators will review the medical records for patients who underwent laparoscopic cholecystectomy.

The patients underwent cholecystectomy using a new technique in approaches to critical safety with recorded video and available follow up data were included.

The patients who had intraoperatively extensive gallbladder adhesion that interfere with the dissection in this area, improper visualization of the cystic duct, patients whose did not operate by this new technique and patients whose have not video record of laparoscopic cholecystectomy will excluded from the study.

DETAILED DESCRIPTION:
Operative procedure:

This technique was different from the ordinary laparoscopic cholecystectomy in the following steps: with the aid of electrocautery Hook, the dissection started first with the peritoneum, which covered both sides of the Hartman pouch, the proximal third of the gallbladder (the area of the gallbladder at its neck), and the proximal part of the cystic duct (the end of the cystic duct which was attached to the gallbladder neck).

With using a grasper for manipulating the Hartman pouch for better dissection of the gallbladder bed. Then gently dissecting the gallbladder from its bed to skeletonize it away from the cystic plate and porta hepatis. The small branches of cystic artery that were dipping in the GB wall were cauterized one by one. This step involved scarification of the cystic artery, and its branches, which necessitated the use of bipolar diathermy.

Now, after dissection of the proximal part of the gallbladder from its bed and scarification of the cystic artery and its branches, the traction applied to the Hartman pouch created an angle between the skeletonized cystic duct and the skeletonized posterior surface of the GB.

Also, this traction creates a dynamic triangle visualized from both the left and right sides according to the traction applied to the Hartman pouch to the right or left and the direction of the angled scope of the camera lens.

From the left-side view, when right traction is applied to the Hartman pouch, it is bound laterally by the skeletonized proximal part of the cystic duct. Superiorly, it is bound by the posterior surface of the proximal part of the skeletonized gallbladder. It was bounded medially by an imaginary line between a point at the junction of the cystic duct with the CBD and a point at the anterior end of the dissected cystic plate (the Madany triangle).

From the right-side view, when left traction was applied on the Hartman pouch, the triangle was bounded by the proximal part of the dissected cystic duct medially. It was bound superiorly by the posterior surface of the proximal third of the skeletonized gallbladder. Laterally, it was bounded by an imaginary line between a point at the junction of the cystic duct with the CBD and another point located at the anterior end of the dissected cystic plate.

A Vicryl (2-0) ligature or a titanium clip was applied to the cystic duct immediately distal to the Hartman pouch after gentle milking of the cystic duct to exclude the presence of stones inside. The GB was removed from the peritoneal cavity with the use of a bag.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute or chronic gall bladder dieses and managed by laparoscopic cholecystectomy.
* Patients undergo laparoscopic cholecystectomy using Madani triangle approaches.

Exclusion Criteria:

* The patients who had intraoperatively extensive gallbladder adhesion.
* Patients managed by open surgical cholecystectomy approaches not laparoscopic.

Ages: 8 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all patients male or female , adult or child underwent laparoscopic cholecystectomy using a new visualized technique Madani triangle
Sampling Method: Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Is the extrahepatic bile duct still intact or injurie. How many patients with the Common bile ducts will injurie? | December 2019 to March 2023
  Is laparoscopic cholecystectomy using Madani triangle technique associated with bile duct injuries or not associated with bile duct injuries or not?

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Abdelmohsen, Lecturer, Principal Investigator — Aswan University
Locations (1):
- Aswan university, Aswān, Aswan Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Madani triangle is a new visualized triangle for laparoscopic cholecystectomy
Supporting Information: Study Protocol
Time Frame: December 2019- March 2023
Access Criteria: Herein, we describe another triangle with a CVS because the dissection and cauterization of the cystic artery are in the area of the proximal part of the cystic duct (CD) at its junction with the gallbladder (GB) neck, away from the common bile duct (CBD) and right hepatic artery. So, the surgical steps are far from the CT and its medial structure boundary.